CLINICAL TRIAL: NCT05221307
Title: Effects of Modified Pilates Training on Hemodynamic Responses in Children With Cerebral Palsy
Brief Title: Effects of Modified Pilates Training on Hemodynamic Responses
Acronym: cp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSU4
Record Dates: First submitted 2022-01-05; First posted 2022-02-02 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy; Physical Inactivity; Gait Disorders in Children; Gait, Spastic
Keywords: Cerebral Palsy; modified pilates exercises; neurodevelopmental therapy; hemodynamic responses
MeSH Terms: conditions — Cerebral Palsy; Sedentary Behavior; Gait Disorders, Neurologic | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The intervention will be rehabilitation methods applied with different exercise trainings, Neurodevelopmental Therapy (NGT-Bobath) will be applied to one group and Modified Pilates Exercises (MPE) (non-invasive) will be applied to the other group.
Who Masked: Investigator
Masking Description: Treatments will be carried out by the same physiotherapist. Evaluations will be made twice, before and after the treatment. All assessments will be made by a different physician physiotherapist who is unfamiliar with the treatment groups. Individuals with CP in the study groups will continue with a blind physiotherapist experienced in pediatric rehabilitation who has completed the training in modified pilates, is certified by The Australian Physiotherapy Pilates Institute (APPI) and has NDT-Bobath certification.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1/Children with cerebral palsy (Experimental): Modified Pilates Exercises (MPEs) will be applied 3 days a week, 45 minutes a day for 8 weeks.
  Interventions: Other: exercises
- 2/children with cerebral palsy (Active Comparator): Traditional Neurodevelopmental Therapy (NGT-Bobath) approach will be applied for 45 minutes a day, 3 days a week for 8 weeks.
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — Group 1 will be given MPEs for 45 minutes, 3 days a week for 8 weeks. In the second group, traditional Neurodevelopmental Treatment (NGT-Bobath) approach will be applied for 45 minutes a day, 3 days a week for 8 weeks. Treatments will be carried out by the same physiotherapist. Evaluations will be made twice, before and after the treatment.

SUMMARY:
Cerebral Palsy (CP) is a non-progressive neurodevelopmental disorder that starts in the early stages of life, causes activity limitation, and consists of movement and posture deficiencies. Children with CP usually have difficulties in mobility, transfer and social participation due to many motor and sensory disorders such as muscle weakness, decreased postural control, balance, spasticity. Core stability maintains posture and provides support for extremity movements by connecting with the deep abdominal muscles, spine, pelvis and shoulder girdle muscles. During reaching, walking and sudden perturbations in the body, the Transversus Abdominus (TrAb) muscle is activated primarily than other trunk and extremity muscles, creating a core stability. Core activity includes not only spinal stability and power generation, but also many upper and lower extremity movements. By focusing on the TrAb muscle with Pilates, the stabilization of the trunk muscles can be increased by creating control thanks to the core stabilization training. In addition, the TrAb muscle works together with the diaphragm muscle, which is the main respiratory muscle. The expected increased respiratory capacity with training may also affect hemodynamic responses.

DETAILED DESCRIPTION:
Children with CP usually have difficulties in mobility, transfer and social participation due to many motor and sensory disorders such as muscle weakness, decreased postural control, balance, spasticity. Abnormal motor patterns and tone, poor trunk control, and postural disorders adversely affect the physical development of these children. Children with CP show deficits in proximal muscle co-contraction and posture stabilization, which leads to limitations in postural reactions and antigravity movements. Dysfunctions are also observed in antisipatory and reactive postural adjustments, and limitations occur especially in upper extremity functions such as walking, reaching, and eating. Although these limitations associated with postural control dysfunctions are known, optimal intervention methods have not yet been determined. Because of these dysfunctions, many individuals with CP have difficulty walking independently, walking on slopes/uneven ground, and performing daily physical functions. Trunk control, which is formed by the activation of the core muscles, is the determinant of postural control, automatic postural reactions, balance, walking and functional activities from the early period.By focusing on the TrAb muscle with Pilates, the stabilization of the trunk muscles can be increased by creating control thanks to the core stabilization training. In addition, the TrAb muscle works together with the diaphragm muscle, which is the main respiratory muscle. The expected increased respiratory capacity with training may also affect hemodynamic responses. Proximal extremity muscles around the hip are also important for maintaining upright posture and maintaining mobility. Studies have shown that hip abductor muscle strength is more associated with gait variables and motor functions in children with CP compared to knee and ankle muscles. Although the importance of this in terms of gait has been determined, studies investigating the activation patterns of trunk and hip muscles during walking of individuals with CP are limited.For this reason, it is thought that pilates training can be applied in terms of muscle strength and postural control in selected individuals with CP who can walk, stand independently, but need to develop some components for controlled movement.Although there are a limited number of studies investigating the effects of modified pilates exercises (MPE) in individuals with CP in different clinical types, their effects on trunk control, core muscle endurance, hemodynamic responses and gait have not been investigated. It is known that most children with CP have significantly lower performance in cardiorespiratory and metabolic tests than their healthy peers.For many of these children, these mobility limitations associated with physical activity adversely affect musculoskeletal and cardiovascular function and increase the risk for secondary medical conditions. Therefore, viable, effective interventions are needed to improve the mobility and cardiorespiratory performance of children with CP. For example, bodyweight supported treadmill training has been used to address these children's walking and fitness goals. However, its routine use in smaller clinics, schools and home settings is often not feasible given the physical requirements associated with helping a child with significant weakness, spasticity or cardiovascular endurance deficiencies keep pace.For this purpose, it is noteworthy that the effects of MPE training targeting the TrAb muscle on gait and hemodynamic responses have not been investigated, especially in children with CP.This study aims to determine the effects of modified pilates exercises (MPE) and traditional neurodevelopmental therapy (NDT-Bobath) on hemodynamic responses in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CP according to Surveillence Of Cerebral Palsy İn Europe (SCPE) criteria
* Can be classified as level I, II or III by GMFCS-E&R [29]
* Children 7-14 years old
* Able to stand up from sitting and walk with or without mobility devices
* No limitation in range of motion in lower extremities and trunk
* Lower extremity spasticity between 1 and 1+ according to the Modified Ashworth (MASH) score
* Individuals with hemiparetic-diparetic CP who can follow verbal commands

Exclusion Criteria:

* Multiple disabilities (hearing, speaking, seeing)
* Congenital cardiorespiratory problem
* Known additional cardiorespiratory disease (asthma, chronic bronchitis, etc.)
* Have taken any special pilates training in the last 6 months
* Not having had any botox/surgery with the lower extremity in the last 6 months

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
6MWT | the change of the 6MWT meter after 8 weeks
  Six minute walk test (6MWT) distance will be recorded as meter.
The Observational Gait Scale (OGS) | change from baseline after 8 weeks
  The Observational Gait Scale was created by developing and modifying the measurement sensitivity of the Physician Rating Scale (PRS). OGS consists of knee position in the middle of the stance phase, first foot contact, foot contact in the middle of the stance phase, time of heel lift, rear foot position in the middle of the stance phase, and support area width. Each leg is evaluated separately and a person with normal gait can get a maximum of 22 points. Higher score indicates better performance.
Sharman's core stability test (PBU=Pressure Biofeedback Unit Test) | change from baseline after 8 weeks
  TrAb muscle strength measurement Sharman's core stability test (PBU=Pressure Biofeedback Unit Test) will be recorded as mm Hg.
Modifiye Beiring Sorensen Test | change from baseline after 8 weeks
  core stabilitiy performance test of Modifiye Beiring Sorensen Test will be recorded as second (s).
Prone Plank Test | change from baseline after 8 weeks
  core stability performance test of Prone Plank Test will be recorded as second (s).
Side Plank Test | change from baseline after 8 weeks
  core stability performance test of Side Plank Test will be recorded as second (s).
Abdominal Fatigue Test | change from baseline after 8 weeks
  core stability performance test of Abdominal Fatigue Test will be recorded as second (s).
Sits Ups Test | change from baseline after 8 weeks
  Sits Ups Test will be recorded as second (s).
Push ups Test | change from baseline after 8 weeks
  core power tests of Push ups Test will be recorded as second (s).
blood pressure (BP) | change of the blood pressure before and after 6MWT on the first day of intervention and after the 8 weeks intervention before and after the 6MWT.
  Both systolic and diastolic blood pressure before and after the 6MWT will be measured and recorded as mmHg.
pulse (P) | change of the pulse before and after 6MWT on the first day of intervention and after the 8 weeks intervention before and after 6MWT.
  pulse before and after the 6MWT will be recorded number.
respiratory rate (RR) | hange of the respiratory rate (RR) before and after 6MWT on the first day of intervention and after the 8 weeks intervention before and after 6MWT.
  respiratory rate (RR) before and after the 6MWT will be recorded as number.

SECONDARY OUTCOMES:
Expanded and revised Gross Motor Function Classification System (GMFCS-E&R) | first day of assessment
  It is a standard classification system used to classify gross motor functions of children with CP. GMFCS-E&R classifies levels I to V. Level I indicates the best and V the worst level of motor function.
Modified Ashworth Scale (MAS) | first day of assessment
  Lower extremity muscle spasticity will be measured. MAS is a method used to determine the severity of spasticity. It is based on the subjective rating of the resistance felt during the examination. The tone felt in these muscles against passive movement is classified as follows; 0: No increase in tone, 1: Slight increase in tone characterized by catching and relaxation or mild resistance at the end of the ROM, 1+: Slight increase in tone characterized by minimal resistance in the remaining ROM (less than half) after capture, 2: Significant tone over most of the ROM increase, but the involved joint can be moved easily, 3: Significant increase in muscle tone, passive movement is difficult, 4: The involved part is rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıguzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University; Bulent Elbasan, Proffessor, Study Director — Gazi University
Locations (1):
- Hatice Adıgüzel, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No